CLINICAL TRIAL: NCT06789835
Title: Automated Quantification of Dental Plaque
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: 3Shape A/S (Industry); National and Kapodistrian University of Athens (Other)
Responsible Party: Sponsor
Other Study IDs: 109/2023
Record Dates: First submitted 2024-12-19; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Fluorescence imaging of disclosed and undisclosed plaque
  Interventions: Device: Fluorescence imaging of disclosed and undisclosed plaque

INTERVENTIONS:
Device: Fluorescence imaging of disclosed and undisclosed plaque — Teeth are imaged using a fluorescence camera/an intraoral scanner before and after plaque disclosure.

SUMMARY:
The study generates data that contribute to the development and validation of an automated approach to full-mouth quantification of dental plaque, based on fluorescence images and intraoral scans of teeth with disclosed and undisclosed plaque.

ELIGIBILITY:
Inclusion Criteria:

Males and females ≥ 18 years old Presence of at least one tooth Anatomically possible to perform intraoral imaging Subjects need to be able to understand and follow instructions, as well as to read and sign the informed consent form

Exclusion Criteria:

History of allergies towards any of the ingredients in the disclosing agents Self-reported serious medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Planimetric plaque index | 1 day
  Plaque area coverage of teeth

SECONDARY OUTCOMES:
Turesky modification of the Quigley and Hein Plaque Index | 1 day
  Plaque coverage of teeth

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Schlafer, DDS, Principal Investigator — University of Aarhus
Locations (1):
- Department of Dentistry and Oral Health, Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to general data protection regulations, individual participant data will not be made available publicly. Summary data will be made available upon publication of the results.